CLINICAL TRIAL: NCT06527209
Title: Chemical and Sensory Characterization of a Drink Based on Coffee and Agave Inulin and Its Effect on Appetite, Dietary Intake, and Biochemical Profile in Subjects With Obesity
Brief Title: Effect of Coffee and Agave Inulin-based Beverage on Appetite in Adults With Obesity.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Livier Nathaly Torres Castillo, Associate Professor B, University of Guadalajara
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CI-02523; 0602-23 HCJIM-2023 (Other: Secretaria de Salud Jalisco)
Record Dates: First submitted 2024-03-01; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Obesity
Keywords: coffee; agave inulin; obesity; ghrelin; GLP-1; PYY; appetite; visual analogue scale; specific sensory satiety; sensory specific desire
MeSH Terms: conditions — Obesity | interventions — Coffee

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to the two interventions separately according to the random assignment sequence corresponding to the crossover design. The interventions consist of a control beverage or a coffee and inulin-based beverage. The beverage will consumed daily 30 minutes before breakfast for two weeks with a two-week washout period.
Who Masked: Participant, Care Provider
Masking Description: In order to minimize implementation biases, participants will be masked, and will not be told whether they are receiving the intervention or the control, to avoid any influence on the data they report on the scales, and the people in charge of administering the intervention will be masked by coding the data to allow the identification of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Active Comparator): Participants receive 350 g of a coffee and agave inulin-based beverage (A) at the fasting state 30 minutes before breakfast for two weeks, and after a two-week washout period, they will receive 350 g of a control beverage (B) at the fasting state, 30 minutes before breakfast for two weeks.
  Interventions: Other: Coffee and agave inulin-based beverage (A); Other: Control beverage (B)
- Sequence BA (Active Comparator): Participants receive 350 g of a control beverage (B) at the fasting state 30 minutes before breakfast for two weeks, and after a two-week washout period, they will receive 350 g of a coffee and agave inulin-based beverage (A) at the fasting state, 30 minutes before breakfast for two weeks.
  Interventions: Other: Coffee and agave inulin-based beverage (A); Other: Control beverage (B)

INTERVENTIONS:
Other: Coffee and agave inulin-based beverage (A) — Intervention beverage:
  134 mL of cold-brew coffee 18 g of agave inulin Total beverage weight: 350 g
  Other Names: Intervention beverage
Other: Control beverage (B) — Control beverage:
  40 mL of cold brew coffee 5.4 g of agave inulin Total beverage weight: 350 g.

SUMMARY:
Nutritional treatment is key in managing obesity; however, the lack of fullness or satiety signals may affect adherence to this treatment. Coffee and inulin consumption, separately, have been shown to increase satiety and GLP-1 concentrations and reduce appetite and energy intake, but they have not been evaluated together. It is necessary to obtain scientific evidence contributing to recommendations for controlling appetite in an obesity context.

Therefore, this study aims to analyze the use of coffee and agave inulin-based beverage consumption on appetite sensations, dietary intake, and ghrelin, GLP-1, and PYY concentrations in adults with obesity.

For that purpose, a double-blind, randomized crossover clinical trial was designed to evaluate the effect of daily consumption, during two weeks, of a coffee and inulin-based beverage compared to a control beverage. Appetite sensations will be analyzed with visual analogue scales, dietary intake with a 3-day self-reporting of food intake, and appetite hormones with ELISA assays. The measurements will be performed in 6 scheduled sessions. In each session, fasting and postprandial appetite variables will be evaluated.

DETAILED DESCRIPTION:
In Mexico, obesity has not ceased to increase since 1988, when it had a prevalence of only 9.5% compared to the 36.1% recorded in 2018, so it is necessary to start acting for the welfare of the Mexican population. In the search for a tool to complement nutritional intervention, we found coffee and inulin. Coffee consumption in our country increases 2% each year and according to data from PROFECO (Procuraduría Federal del Consumidor), 85% of Mexicans beverage one to three cups a day.

Agave tequilana Weber, a blue variety, is the most widely cultivated of the 117 species of agaves native to Mexico, a variety that is an important source of inulin.

Based on previous research, these two products of the Mexican countryside have been shown to provide health benefits, each in their own right. In the case of coffee, it has been shown to improve endurance and exercise capacity, has antioxidant capacity, has been associated with a lower risk of Parkinson's and Alzheimer's disease, and several studies report a hepatoprotective effect. Regarding appetite control and weight loss, there is still great controversy within the scientific community about its effects, especially due to the lack of randomized clinical trials. Inulin has been shown to improve intestinal transit, lower LDL cholesterol, and be an important prebiotic for the intestinal microbiota. However, its relationship with appetite control is unclear. These effects on regulating appetite processes such as hunger and satiety have been studied in other countries, but not in Mexico, and much less so using inulin from agave tequilana Weber.

Part of this project is to design a beverage based on coffee and agave inulin that provides health benefits, but that is also to the taste and consumption preferences of the population so that it can be easily included as part of their regular diet, that has a low energy content and also contains the necessary amount of bioactive compounds that have proven to have beneficial effects on health, and that could have an improvement in appetite control, according to the background that has been reported. All this is supported by the clinical trial proposed in this research project. In addition, this beverage could represent an option of an accessible food that could be a healthy alternative to sugary beverages with low fiber intake that are consumed with great demand in our country.

Objective: To evaluate the chemical and sensory characteristics of coffee and agave inulin-based beverages and their effects on appetite, dietary intake, and biochemical profiles in subjects with obesity.

Type of study: Double-blind, randomized crossover clinical trial

All participants will be assigned to two interventions separately, according to the random assignment sequence corresponding to the crossover design.

The interventions consist of consuming a beverage (intervention or placebo) daily 30 minutes before breakfast for two weeks, with an intermediate washout period of 2 weeks between each treatment. Participants will be assigned randomly to the sequence AB (intervention beverage/placebo) or BA (placebo/intervention beverage) by generating a table of random numbers in the SPSS software.

Subjects who attend the Bariatric and Metabolic Surgery Unit of the Nuevo Hospital Civil de Guadalajara "Dr. Juan I. Menchaca" and who meet the selection criteria. Subjects attend six sessions, one each week.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 25 to 55 years of age
* BMI ≥ 30 and <35 kg/m2
* Habitual coffee consumption (1 - 3 cups of 240 ml of coffee per day)
* Willingness to stop consuming food and/or supplements with coffee, caffeine and/or inulin during the study with the exception of the intervention
* Availability of time in the mornings
* Residents of the Guadalajara Metropolitan Area
* Signed informed consent form

Exclusion Criteria:

* Hypersensitivity or intolerance to coffee or inulin
* Allergy or intolerance to any of the test foods
* Current or within the last 6 months use of weight-loss or appetite altering medications appetite altering medications
* Diagnosis of diabetes, hypertension or any heart disease, thyroid disease, infectious disease (COVID-19, flu, etc.), digestive or inflammatory bowel disease or dysgeusia
* Smoking
* Women who are pregnant, want to become pregnant, or are breastfeeding
* Peri-menopausal or menopausal women
* Who are on any dietary regimen for weight loss
* Currently or within the last 12 months participated in another study
* Consumption of prebiotics or probiotics in the last three months
* Incomplete data and/or measurements
* Lack of expected compliance (drinking at least 5 of the 7 days of each week is considered compliance).
* Individuals who decide to leave the study

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the subjective appetite sensations when consuming the intervention beverage vs. the control beverage. | Basally and two weeks after taking the intervention beverage. Basally and two weeks after taking the control beverage. In total, on four occasions. And on each occasion, they will be measured at times -30, 0 (beverage consumption), 30, and 60 minutes.
  The subjective appetite sensations are measured with the visual analogue scales (VAS). VAS are made up of lines, usually 100 mm long, with the term "None" or "Not at all" at one end and "Yes, very much" at the other end. or "As much as I have never felt." The subject marks a point between these two extremes, and the quantification is done by measuring the distance from the left end of the line to the mark to which a score is given. These scales are validated and reproducible instruments. The VAS assesses hunger, fullness, satiety, desire to eat, prospective consumption, and the desire for sweet, salty, fatty, and savory food.
Comparison of acylated ghrelin concentrations when consuming the intervention drink vs. the control drink. | Basally and two weeks after taking the intervention drink. Basally and two weeks after taking the control drink. In total, on four occasions. And on each occasion, it will be measure at -30 and 30 minutes after consumption of the beverage
  Ghrelin is determined by an enzyme-linked immunosorbent assay (ELISA) kit. The kit is based on a double antibody sandwich technique. The plate wells are coated with a monoclonal antibody specific to the C-terminal region of ghrelin. This antibody will bind to any ghrelin introduced into the wells, whether standard or sample. In addition, the acetylcholinesterase (AChE)-Fab (Marker) conjugate that recognizes the N-terminal region of ghrelin is introduced into the wells. The two antibodies thus form a sandwich by binding to different parts of the acylated ghrelin. The AChE marker acts on the substrate solution (Ellman's reagent) to generate a yellow compound with strong absorption at 405 or 414 nm. The intensity of the color, measured spectrophotometrically, is directly proportional to the amount of acylated (human) ghrelin. For this purpose, the plate will be read on a Thermo Scientific Multiskan Sky spectrophotometer.
Comparison of the glucagon-like peptide 1 (GLP-1) levels when consuming the intervention beverage vs. the control beverage. | Basally and two weeks after taking the intervention drink. Basally and two weeks after taking the control drink. In total, on four occasions. And on each occasion, it will be measured at times -30 and 30 minutes after consumption of the beverage.
  The determination of GLP-1 levels is done by an enzyme immunoassay (EIA) kit (Biovendor Cat. No. YK160). This EIA kit is used to determine human GLP-1 in plasma samples quantitatively. Its sensitive quantification and high specificity characterize the kit. In addition, it is not influenced by the other constituents in the samples.
  This EIA kit for determining rat/mouse/human GLP-1 in plasma samples is based on a competitive enzyme immunoassay using a combination of highly specific antibodies to GLP-1, amide, and biotin-avidin affinity system. To the well of the plate coated with goat anti-rabbit IgG, GLP-1 standard or samples labeled antigen and GLP-1 antibodies are added for competitive immunoreaction. After incubation and plate washing, horse radish peroxidase (HRP) labeled streptoavidin (SA) is added to form HRP labeled SA-biotinylated GLP-1 - antibody complex on the surface of the wells.
Comparison of the PYY levels when consuming the intervention beverage vs. the control beverage. | Basally and two weeks after taking the intervention drink. Basally and two weeks after taking the control drink. In total, on four occasions. And on each occasion, it will be measured at times -30 and 30 minutes after the beverage consumption.
  The determination of PYY levels is done by an enzyme immunoassay (EIA) kit (Biovendor Cat. No. YK080). This EIA kit is used to determine human PYY in serum and plasma samples quantitatively. Its sensitive quantification and high specificity characterize the kit. In addition, it is not influenced by other components in samples. This determination is based on a competitive enzyme immunoassay using a combination of highly specific antibodies to the human PYY and a biotin-avidin affinity system. To the wells of plate coated with rabbit anti-human PYY antibody, standard or samples, labeled antigens are added for competitive immunoreaction. After incubation and plate washing, horse radish peroxidase (HRP) labeled streptoavidin (SA) is added to form HRP labeled streptoavidin-biotinylated antigen-antibody.
Comparison of dietary intake when consuming the intervention beverage vs. the control beverage. | 3 days, being a weekday, a weekend day, and the day before the session
  Participants will complete six 24-hour reminders: two weekend days, three weekdays, and the day before they finish the first sequence. Participants will complete six 24-hour reminders: two weekend days, three weekdays, and the day before they finish the second sequence. The diet analysis will be carried out on the Nutritionist ProTM software.
Comparison of liking and wanting for specific foods when consuming the intervention beverage vs. the control beverage. | Basally and two weeks after taking the intervention beverage. Basally and two weeks after taking the control beverage. In total, on four occasions. And on each occasion, they will be measured at times -30, 0 (beverage consumption), 30, and 60 minutes.
  The specific sensory satiety is measured with the visual analogue scales (VAS). VAS are made up of lines, usually 100 mm long, with the term "None" or "Not at all" at one end and "Yes, very much" at the other end. or "As much as I have never felt." The subject marks a point between these two extremes, and the quantification is done by measuring the distance from the left end of the line to the mark to which a score is given. These scales are validated and reproducible instruments. The VAS assesses liking and wanting, which is the motivational aspect of appetite or inclination to consume a specific food.
Comparison of specific sensory desire when consuming the intervention beverage vs. the control beverage. | Basally and two weeks after taking the intervention drink. Basally and two weeks after taking the control drink. In total, on four occasions. And on each occasion, they will be measured at -30, 0 (beverage consumption), 30, 30 and 60 minutes.
  The specific sensory desire is measured with the visual analogue scales (VAS). VAS are made up of lines, usually 100 mm long, with the term "None" or "Not at all" at one end and "Yes, very much" at the other end. or "As much as I have never felt." The subject marks a point between these two extremes, and the quantification is done by measuring the distance from the left end of the line to the mark to which a score is given. These scales are validated and reproducible instruments. Using these VAS, participants will be instructed to rate their desire to eat something sweet, salty, sour, bitter, fatty, and spicy.
Comparison of food choice when consuming the intervention beverage vs. the control beverage. | Basally and two weeks after taking the intervention drink. Basally and two weeks after taking the control drink. In total, on four occasions. And on each occasion, it will be measured at 60 minutes.
  The evaluation of food choice consists of serving food samples with certain sensory properties: (1) peach in syrup as sweet, (2) green apple with lemon drops as sour, (3) cracker as salty, (4) cocoa nibs as bitter, (5) jalapeño bell pepper as spicy, (6) avocado as "fatty", (7) chocolate sandwich cookie with vanilla-flavored filling as an ultra-processed sweet food, (8) cheese-flavored totopo as ultra-processed salty food, and (9) a sample of the coffee and inulin-based beverage from either the intervention or control. Participants will be instructed to choose the 3 test foods they would eat the most and the one they would eat the least at that time.

SECONDARY OUTCOMES:
Comparison of biochemical profile when consuming the intervention beverage vs. the control beverage. | Initially and two weeks after taking the intervention drink. Basally and two weeks after taking the control drink. In total, on four occasions. And on each occasion, it will be measured fasting and 30 minutes after consumption of the beverage
  The concentration of glucose, triglycerides, total cholesterol, and high-density lipoprotein cholesterol (HDL-c) was determined with a dry chemistry analyzer Vitros 350 Chemistry (Ortho-Clinical Diagnostics, Johnson & Johnson Services Inc., Rochester, NY, USA). Low-density lipoprotein cholesterol (LDL-c) was calculated with the Friedewald formula, except when triglyceride levels were greater than 400 mg/dL (5). Very-low-density lipoprotein cholesterol (VLDL-c) was calculated as total cholesterol minus the sum of LDL-c + HDL-c

CONTACTS AND LOCATIONS:
Overall Officials: Livier N Torres, Ph.D, Study Director — University of Guadalajara
Locations (1):
- Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT06527209/Prot_000.pdf
  • Informed Consent Form (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT06527209/ICF_001.pdf